CLINICAL TRIAL: NCT00743470
Title: A Comparison of the Bioavailability of Rifabutin With and Without Lopinavir/Ritonavir in Healthy Adult Subjects
Brief Title: A Bioavailability Study of Rifabutin and Lopinavir/Ritonavir in Healthy Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Daniel Cohen, MD/Study Medical Director, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-457
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-09

CONDITIONS: HIV; Tuberculosis
Keywords: HIV co-infected with tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Lopinavir; lopinavir-ritonavir drug combination; Rifabutin

ARMS (2):
- A, B (Experimental): Group 1 receives regimen A and B. A: Healthy volunteers, receiving one 150 mg rifabutin QD alone. B: Healthy volunteers, receiving 150 mg rifabutin QD+ two lopinavir/ritonavir 200/50 mg tablets BID.
  Interventions: Drug: lopinavir/ritonavir; Drug: rifabutin
- C (Experimental): Group 2 receives regimen C. C: 150 mg rifabutin QD+ two lopinavir/ritonavir 200/50 mg tablets BID.
  Interventions: Drug: lopinavir/ritonavir; Drug: rifabutin

INTERVENTIONS:
Drug: lopinavir/ritonavir — lopinavir/ritonavir tablet; see arm for intervention description
  Other Names: ABT-378; Kaletra
Drug: rifabutin — rifabutin capsule; see arms for intervention description

SUMMARY:
The purpose of this study is to study the safety, tolerability and pharmacokinetics of rifabutin dosing with lopinavir/ritonavir tablets in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult Male or Female 18-55 yrs.
* Subject has provided written consent.
* Subject is in general good health.
* If female, subject is postmenopausal.
* If female, subject is not pregnant and is not breast-feeding.
* Subject must use birth control methods or be surgically sterile.

Exclusion Criteria:

* Subject is HAV-IgM, HBsAg or HIV Ab positive.
* Positive screen for drugs of abuse, alcohol, or smoking.
* Cannot be on any medication, including over the counter drugs.
* Cannot have previous history of alcohol or drug abuse.
* Cannot have history of any major diseases or disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Analysis of pharmacokinetic variables will be computed for each sampling time and each parameter. | Approximately 0.5 - 1 month
Analysis of safety measures including but not limited to tabulation of adverse events, physical exam, clinical lab results (include chemistry, hematology and urine) and vital signs. | Approximately 0.5 - 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Angela Nilius, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 11441, Waukegan, Illinois, United States